CLINICAL TRIAL: NCT03673631
Title: Evaluation of Oxygenation Methods and Non-invasive Ventilatory Support in Patients With Acute Respiratory Failure for Whom a Do-not Intubate Order Was Taken: Prospective Observational Study
Brief Title: Oxygenation Methods and Non-invasive Ventilation in Patients With Acute Respiratory Failure and a do Not Intubate Order
Acronym: OXYPAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OXY-PAL
Record Dates: First submitted 2018-08-02; First posted 2018-09-17 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Acute Respiratory Failure; Cancer; Hematologic Malignancy; Cardiac Insufficiency; Chronic Respiratory Insufficiency
Keywords: non-invasive ventilation; nasal high flow humidified canula oxygenation; palliative; acute respiratory failure; withholding therapies; withdrawing therapies
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NFHC-O2 Group: NFHC-O2 therapy alone with gas flow at least 40L/min,
  Interventions: Device: NFHC-O2
- NIV/Standard-O2 Group: NIV sessions with at least 30% FiO2 and standard oxygen therapy
  Interventions: Device: NIV
- NFHC-O2/NIV Group: combination of NIV sessions and NFHC-O2 therapy,
  Interventions: Device: NIV; Device: NFHC-O2

INTERVENTIONS:
Device: NIV — NIV setting: minimal FiO2 0.3; tidal volume 6-8ml/kg (theoretical body weight)
  Groups: NFHC-O2/NIV Group; NIV/Standard-O2 Group
Device: NFHC-O2 — NFHC-O2 setting: minimal FiO2 0.3; minimal flow 40l/min
  Groups: NFHC-O2 Group; NFHC-O2/NIV Group

SUMMARY:
ICU care of patients considered "palliative" but without contraindications to admission to intensive care, for whom a do-not intubate order decision was made upon admission represents a particular target for non-invasive oxygenation techniques. The benefits of non invasive ventilation (NIV) in this population are debated especially in cancer patients. The more recently used nasal humidified high flux canula oxygenation (HFNC) therapy may have benefits over NIV in these patients. It is supposed to have better tolerance and could allow better compliance and thus higher efficiency. These potential benefits are major for such a population for which tolerance and symptomatic relief are priority goals

DETAILED DESCRIPTION:
Observational prospective multicenter study Primary outcome: To analyze the efficacy and tolerance of NIV and HFNC in patients admitted to intensive care unit, or intermediate catre unit for acute respiratory insufficiency for whom a a do-not intubate order decision was taken upon admission or after extubation if the patient initially received mechanical ventilation.

Secondary outcomes: To analyze the efficacy and tolerance of NIV and HFNC according to the following reason for ICU admission: chronic obstructive pneumopathy decompensated COPD, severe heart failure, evolutive cancer or hematologic malignancy; to analyze tolerance and acceptability of different techniques; to analyze the duration of the oxygenation methods use; to analyze the modalities of eventual withdrawing life support therapies and the associated sedative and opioid treatments; to analyze the satisfaction for the use of the non invasive technique by the relatives and the caregivers; to analyze mortality at D28 and D90 and quality of life at 3 and 6 months in surviving patients

ELIGIBILITY:
Inclusion Criteria:

* acute respiratory failure defined by respiratory rate>25/min and or hypoxemia (sPO2 <92% with O2 >3l/min)
* admission in ICU or intermediate care unit
* decision to not intubate the patient or to not re-intubate the patient
* indication to NIV or HFNC-O2
* French social security affiliation

Exclusion Criteria:

* refusal to participate
* legal protection
* pregnancy
* prophylactic treatment by VNI or HFNC-O2 after extubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * patient admitted in ICU or intermediate care with decision of a do-not intubate order on admission or after extubation (for patients receiving invasive mechanical ventilation)
  * with acute respiratory failure criteria (respiratory rate >25/min; contraction of accessory respiratory muscles or hypoxemia requiering > 3L/min O2 to obtain SpO2 >92%)
  * and having indication for NIV or HFNC-O2
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Survival at day 14 | day 14
  Survival at day 14 in patients weaned from NIV and or HNFC-O2

SECONDARY OUTCOMES:
Clinical respiratory parameters evolution | day 1, day 2, day 3
  respiratory rate improvement will be assessed by a decrease of respiratory rate below 20/min
Oxygenation parameters evolution | day 1, day 2, day 3
  sPO2 (oxygen saturation) expressed in % improvement will be assessed by an increase above 92%
tolerance of technique of oxygenation | day 1, day 2, day 3
  tolerance will be assessed by comfort visual analogic scale from 1 worse tolerance to 10 very good tolerance; improvement defined as a 20% decrease of the value
evolution of quality of life | on admission and after 3 and 6 months after ICU stay
  quality of life will be measured by the EuroQuality of life 5D score (EQ5D) recording 5 subscore (mobility, autonomy, ability to perform current activities, pain, anxety/depression); the value of each is from 1 to 3 points; total score is the sum of the 5 subscores with a minimal score of 5 and a maximal score of 15. The baseline score will be recorded after admission in the ICU and reflects the patient's quality of life just before his or her admission. After 3 and 6 months, a higher value of the score will represent a worse outcome.
Acceptation of the non invasive technique | day 14
  tolerance defined by the absence of refusal to continue the technique (NIV or HNFC O2) by the patient
mortality day 28 | day 28
  percentage of patients deceased at day 28 whatever the cause of death

CONTACTS AND LOCATIONS:
Overall Officials: René ROBERT, MD,PhD, Study Director — Poitiers University Hospital
Locations (1):
- Chu de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robert R, Frasca D, Badin J, Girault C, Guitton C, Djibre M, Beuret P, Reignier J, Benzekri-Llefevre D, Demiri S, Rahmani H, Argaud LA, I'her E, Ehrmann S, Lesieur O, Kuteifan K, Thouy F, Federici L, Thevenin D, Contou D, Terzi N, Nseir S, Thyrault M, Vinsonneau C, Audibert J, Masse J, Boyer A, Guidet B, Chelha R, Quenot JP, Piton G, Aissaoui N, Thille AW, Frat JP. Comparison of high-flow nasal oxygen therapy and non-invasive ventilation in ICU patients with acute respiratory failure and a do-not-intubate orders: a multicentre prospective study OXYPAL. BMJ Open. 2021 Feb 12;11(2):e045659. doi: 10.1136/bmjopen-2020-045659. PMID 33579774